CLINICAL TRIAL: NCT03927690
Title: A Randomized, Active-controlled, Patient and Investigator-masked, Multiple Dose Proof-of-concept Study of Intravitreal LKA651 in Patients With Diabetic Macular Edema
Brief Title: Multiple Dose Safety and Efficacy of LKA651 in Patients With Diabetic Macular Edema
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CLKA651X2202; 2018-000031-28 (EudraCT Number)
Record Dates: First submitted 2019-04-23; First posted 2019-04-25 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Edema
Keywords: Macular degeneration; age-related macular degeneration (ARMD); vision loss; macula damage; retina damage; dry macular degeneration; wet macular degeneration; AMD; diabetic macular edema; DME; neovascular age-related macular degeneration; nAMD; retinal vein occlusion; RVO; Diabetic Macular edema (DME); macular edema; diabetic retinopathy; LKA651; Lucentis
MeSH Terms: conditions — Macular Degeneration; Vision Disorders; Geographic Atrophy; Wet Macular Degeneration; Retinal Vein Occlusion; Macular Edema; Diabetic Retinopathy | interventions — Ranibizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- LKA651 (Experimental): LKA651 Intravitreal injection
  Interventions: Drug: LKA651
- LKA651 + Lucentis (Experimental): LKA651 + Lucentis Intravitreal injection
  Interventions: Drug: LKA651; Drug: Lucentis
- Lucentis (Active Comparator): Lucentis Intravitreal injection
  Interventions: Drug: Lucentis

INTERVENTIONS:
Drug: LKA651 — LKA651 5 mg Intravitreal injection, every 4 weeks for 12 weeks in the treatment phase
  Arms: LKA651; LKA651 + Lucentis
Drug: Lucentis — Lucentis 0.3 mg (U.S. sites) or 0.5 mg (ex U.S. sites) Intravitreal injection, every 4 weeks for 12 weeks in the treatment phase
  Arms: LKA651 + Lucentis; Lucentis

SUMMARY:
The primary objectives of this study were to evaluate the safety and efficacy of LKA651 in patients with macular edema from diabetic macular edema (DME),

DETAILED DESCRIPTION:
This study was a 3-arm, parallel group, randomized, patient- and investigator-masked trial planned in 90 patients with Diabetic macular edema (DME). The study consisted of a screening period of 60 days, main study (12 weeks), and an extension period (12 weeks). The study was stratified such that sentinel safety cohorts were first enrolled to test the safety of the combination of LKA651 and Lucentis before proceeding with further patient randomization. After determination of safety from Day 15 data from each sentinel cohort, patients were enrolled into 1 of 3 arms: LKA651 monotherapy, LKA651 plus Lucentis, and Lucentis monotherapy. Every patient was dosed 3 times in 4 week intervals in the treatment phase and was then followed up for an extension phase of an additional 12 weeks during which Lucentis was allowed to be administered as rescue at the discretion of the Investigator. No predefined rescue criteria were outlined as guidance.

ELIGIBILITY:
Inclusion Criteria

* Written informed consent must be obtained before any assessment is performed.
* Male and female patients age 18 to 85 years of age inclusive at screening
* Presence of type I or type II diabetes mellitus
* The Early Treatment Diabetic Retinopathy Study (ETDRS) letter score in the study eye must be between 24 and 70 letters (approximate Snellen equivalent of 20/40-20/320). The non-study eye (fellow eye) should be ≥34 letters or better (approximate Snellen equivalent of 20/200) at screening
* Presence of Diabetic macular edema (DME) in the study eye, with decrease in vision due to foveal thickening of central macular thickness ≥ 320 µm in the central subfield, as assessed on Spectral domain optical coherence tomography (SD-OCT) and confirmed by the central reading center at screening
* Sufficiently clear ocular media and adequate pupil dilation in the study eye to permit fundus photographs of adequate clarity to measure diameters of retinal arteries and veins at screening

Exclusion criteria

* Patient with history of intravitreal (IVT) anti-vascular endothelial growth factor (VEGF) treatment in the study eye <90 days from baseline
* Patient with history of intraocular corticosteroids including dexamethasone intravitreal implants during the 6 month period prior to baseline. Any prior use of fluocinolone acetonide intravitreal implant (Iluvien) is prohibited regardless of timing
* Laser photocoagulation (macular or panretinal) in the study eye during the 3-month period prior to baseline.
* High risk proliferative diabetic retinopathy
* Patients, with type 1 or type 2 diabetes who have a hemoglobin A1C ≥ 12% at screening.
* Any progressive disease of the retina in the study eye (e.g. uveitis,rod-cone dystrophy) or optic nerve
* Area of macular retinal ischemia (as measured by the foveal avascular zone) ≥ 1000 μm.
* Active intraocular inflammation (graded as trace or above) or active intraocular infection in either eye.
* Current diagnosis of or laboratory evidence for anemia, defined as a hemoglobin <10 g/dL for women and <11 g/dL for men.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2019-05-24 (Actual); Primary Completion 2022-06-17 (Actual); Study Completion 2022-08-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (20):
- United States (7):
  - Novartis Investigative Site, Beverly Hills, California
  - Novartis Investigative Site, Rancho Cordova, California
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, ‘Aiea, Hawaii
  - Novartis Investigative Site, Boston, Massachusetts
  - Novartis Investigative Site, Austin, Texas
  - Novartis Investigative Site, San Antonio, Texas
- Germany (5):
  - Novartis Investigative Site, Berlin
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hanover
  - Novartis Investigative Site, Münster
  - Novartis Investigative Site, Tübingen
- Novartis Investigative Site, Arecibo, Puerto Rico
- Spain (5):
  - Novartis Investigative Site, Seville, Andalusia
  - Novartis Investigative Site, Sant Cugat del Vallès, Catalonia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Córdoba
  - Novartis Investigative Site, Zaragoza
- Turkey (Türkiye) (2):
  - Novartis Investigative Site, Ankara
  - Novartis Investigative Site, Kocaeli

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: Patient Lay Trial Summary — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=1566

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The study population consisted of male and female patients with DME, who were 18 to 85 years of age at screening, and who were either treatment naive or experienced i.e. had been treated with anti VEGF therapy > 90 days before baseline.
Groups:
- LKA651: LKA651 5 mg Intravitreal injection, every 4 weeks for a total of 3 doses in the treatment phase
- LKA651 + Lucentis: LKA651 1 mg + Lucentis 0.3 mg (U.S. sites) or 0.5 mg (ex U.S. sites) Intravitreal injection, every 4 weeks for a total of 3 doses in the treatment phase
- Lucentis: Lucentis 0.3 mg (U.S. sites) or 0.5 mg (ex U.S. sites) Intravitreal injection, every 4 weeks for a total of 3 doses in the treatment phase
Period: Overall Study
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Started | 28 | 30 | 33
Completed | 21 | 27 | 31
Not Completed | 7 | 3 | 2
Not completed — Withdrawal by Subject | 3 | 1 | 1
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis | Total
Number analyzed (Participants) | 28 | 30 | 33 | 91
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.6 (8.58) | 63.8 (8.18) | 61.2 (9.02) | 62.2 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 10 | 32
  Male | 19 | 17 | 23 | 59
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 2 | 1 | 0 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 3 | 0 | 0 | 3
  White | 23 | 27 | 32 | 82
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events
Description: An AE is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation patient.
  The severity of the AEs (mild, moderate, severe) was based on the Common Terminology Criteria for Adverse Events (CTCAE).
  Number of participants in each category is reported in the table. A participant who falls multiple times in one category is counted only once.
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 12 weeks post treatment, up to a maximum timeframe of approximately 24 weeks (approximately 168 days).
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 28 | 30 | 33
Participants
  AEs, Patients with AEs | 20 | 16 | 19
  AEs of mild intensity | 16 | 15 | 19
  AEs of moderate intensity | 8 | 6 | 3
  AEs of severe intensity | 4 | 2 | 1
  Study drug-related AEs | 2 | 1 | 2
  Serious AEs | 3 | 4 | 1
  AEs leading to discontinuation of study treatment | 1 | 0 | 0
  Study-drug related AEs leading to discontinuation of study treatment | 1 | 0 | 0
  Non-serious AEs | 20 | 16 | 19

2. Primary Outcome: Number of Participants With Ocular Adverse Events by Preferred Term in Study Eye
Description: An AE is any untoward medical occurrence (e.g., any unfavorable and unintended sign [including abnormal laboratory findings], symptom or disease) in a patient or clinical investigation patient.
Time Frame: as for outcome 1
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 28 | 30 | 33
Participants
  Patients with at least one ocular AE in study eye | 11 | 7 | 9
  Conjunctival haemorrhage | 1 | 4 | 2
  Diabetic retinal oedema | 2 | 1 | 2
  Diabetic retinopathy | 1 | 1 | 1
  Visual acuity reduced | 3 | 0 | 0
  Vitreous haemorrhage | 1 | 0 | 2
  Dry eye | 0 | 1 | 1
  Macular oedema | 2 | 0 | 0
  Ocular hypertension | 2 | 0 | 0
  Abnormal sensation in eye | 0 | 0 | 1
  Anterior chamber flare | 0 | 1 | 0
  Corneal erosion | 1 | 0 | 0
  Cystoid macular oedema | 1 | 0 | 0
  Dacryostenosis acquired | 1 | 0 | 0
  Eye pain | 1 | 0 | 0
  Eyelids pruritus | 0 | 0 | 1
  Lenticular opacities | 0 | 0 | 1
  Punctate keratitis | 0 | 1 | 0
  Retinal cyst | 1 | 0 | 0
  Retinal detachment | 1 | 0 | 0
  Retinal exudates | 1 | 0 | 0
  Retinal haemorrhage | 1 | 0 | 0
  Vitreoretinal traction syndrome | 0 | 0 | 1

3. Primary Outcome: Number of Participants With Non-ocular Adverse Events (>=2%)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 28 | 30 | 33
Participants | 16 | 15 | 14

4. Primary Outcome: Intraocular Pressure (IOP) in Study Eye
Description: Intraocular pressure was measured per the study site's regular practice.
Time Frame: Screening, and Day 85
Population: Safety analysis set
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 28 | 30 | 33
mmHg
  Screening | 15.1 (3.20) | 14.9 (3.44) | 15.5 (2.88)
  Day 85: number analyzed (Participants) | 24 | 28 | 31
  Day 85 | 15.5 (3.56) | 15.6 (3.67) | 15.2 (3.79)

5. Primary Outcome: Best Corrected Visual Acuity (BCVA) by Early Treatment Diabetic Retinopathy Study (ETDRS) Visual Acuity Charts in Study Eye
Description: BCVA was assessed using Early Treatment Diabetic Retinopathy Study (ETDRS) visual acuity testing charts.
  Visual function of the study eye was assessed using the ETDRS protocol.
  BCVA in study eye was analyzed with a mixed model for repeated measures. The model included treatment, visit, and the treatment by visit interaction as independent variables. An unstructured residual covariance structure was used. Baseline BCVA value and treatment naïve and treatment experienced variable were used as covariates.
  Min and max possible scores are 0-100 respectively. A higher score represents better visual functioning.
Time Frame: Days 2, 8, 15, 29, 43, 57, and 85
Population: Pharmacodynamic analysis set - Participants with a valid measure and without a protocol deviation that would have an impact on the outcome measure.
Measure: Mean (90% Confidence Interval); unit: Scores on a scale
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 25 | 28 | 32
Scores on a scale
  Day 2: number analyzed (Participants) | 6 | 17 | 10
  Day 2 | 61.5 [58.6 to 64.4] | 64.4 [62.3 to 66.6] | 64.1 [61.8 to 66.5]
  Day 8: number analyzed (Participants) | 6 | 16 | 10
  Day 8 | 65.2 [61.7 to 68.7] | 68.6 [66.1 to 71.2] | 66.2 [63.4 to 69.0]
  Day 15: number analyzed (Participants) | 6 | 16 | 10
  Day 15 | 65.9 [62.4 to 69.4] | 68.6 [65.8 to 71.4] | 68.4 [65.4 to 71.3]
  Day 29 | 65.5 [62.6 to 68.4] | 68.2 [65.3 to 71.0] | 68.5 [65.9 to 71.1]
  Day 43: number analyzed (Participants) | 5 | 16 | 8
  Day 43 | 67.8 [64.4 to 71.1] | 70.4 [67.6 to 73.3] | 69.1 [66.2 to 71.9]
  Day 57: number analyzed (Participants) | 24 | 27 | 31
  Day 57 | 67.6 [64.7 to 70.5] | 71.5 [68.6 to 74.4] | 70.0 [67.4 to 72.6]
  Day 85: number analyzed (Participants) | 23 | 27 | 31
  Day 85 | 67.8 [64.8 to 70.9] | 72.5 [69.5 to 75.4] | 70.5 [67.8 to 73.2]
Statistical Analysis 1: Comparison: LKA651 vs Lucentis; Day 2; Test type: Superiority; p = 0.887, Mixed model repeated measures analysis; Difference (Test vs Reference) = -2.6, 90% CI 2-sided [-6.2 to 1.0] — Comparison of model-based mean estimates
Statistical Analysis 2: Comparison: LKA651 + Lucentis vs Lucentis; Day 2; Test type: Superiority; p = 0.431, Mixed model repeated measures analysis; Difference (Test vs Reference) = 0.3, 90% CI 2-sided [-2.6 to 3.2] — Comparison of model-based mean estimates
Statistical Analysis 3: Comparison: LKA651 vs Lucentis; Day 8; Test type: Superiority; p = 0.647, Mixed model repeated measures analysis; Difference (Test vs Reference) = -1.0, 90% CI 2-sided [-5.4 to 3.4] — Comparison of model-based mean estimates
Statistical Analysis 4: Comparison: LKA651 + Lucentis vs Lucentis; Day 8; Test type: Superiority; p = 0.130, Mixed model repeated measures analysis; Difference (Test vs Reference) = 2.4, 90% CI 2-sided [-1.1 to 6.0] — Comparison of model-based mean estimates
Statistical Analysis 5: Comparison: LKA651 vs Lucentis; Day 15; Test type: Superiority; p = 0.818, Mixed model repeated measures analysis; Difference (Test vs Reference) = -2.5, 90% CI 2-sided [-6.9 to 2.0] — Comparison of model-based mean estimates
Statistical Analysis 6: Comparison: LKA651 + Lucentis vs Lucentis; Day 15; Test type: Superiority; p = 0.457, Mixed model repeated measures analysis; Difference (Test vs Reference) = 0.3, 90% CI 2-sided [-3.6 to 4.1] — Comparison of model-based mean estimates
Statistical Analysis 7: Comparison: LKA651 vs Lucentis; Day 29; Test type: Superiority; p = 0.906, Mixed model repeated measures analysis; Difference (Test vs Reference) = -3.1, 90% CI 2-sided [-6.9 to 0.8] — Comparison of model-based mean estimates
Statistical Analysis 8: Comparison: LKA651 + Lucentis vs Lucentis; Day 29; Test type: Superiority; p = 0.566, Mixed model repeated measures analysis; Difference (Test vs Reference) = -0.4, 90% CI 2-sided [-4.1 to 3.3] — Comparison of model-based mean estimates
Statistical Analysis 9: Comparison: LKA651 vs Lucentis; Day 43; Test type: Superiority; p = 0.686, Mixed model repeated measures analysis; Difference (Test vs Reference) = -1.3, 90% CI 2-sided [-5.6 to 3.1] — Comparison of model-based mean estimates
Statistical Analysis 10: Comparison: LKA651 + Lucentis vs Lucentis; Day 43; Test type: Superiority; p = 0.280, Mixed model repeated measures analysis; Difference (Test vs Reference) = 1.4, 90% CI 2-sided [-2.5 to 5.2] — Comparison of model-based mean estimates
Statistical Analysis 11: Comparison: LKA651 vs Lucentis; Day 57; Test type: Superiority; p = 0.849, Mixed model repeated measures analysis; Difference (Test vs Reference) = -2.4, 90% CI 2-sided [-6.3 to 1.4] — Comparison of model-based mean estimates
Statistical Analysis 12: Comparison: LKA651 + Lucentis vs Lucentis; Day 57; Test type: Superiority; p = 0.254, Mixed model repeated measures analysis; Difference (Test vs Reference) = 1.5, 90% CI 2-sided [-2.2 to 5.2] — Comparison of model-based mean estimates
Statistical Analysis 13: Comparison: LKA651 vs Lucentis; Day 85; Test type: Superiority; p = 0.866, Mixed model repeated measures analysis; Difference (Test vs Reference) = -2.7, 90% CI 2-sided [-6.6 to 1.3] — Comparison of model-based mean estimates
Statistical Analysis 14: Comparison: LKA651 + Lucentis vs Lucentis; Day 85; Test type: Superiority; p = 0.198, Mixed model repeated measures analysis; Difference (Test vs Reference) = 2.0, 90% CI 2-sided [-1.9 to 5.8] — Comparison of model-based mean estimates

6. Primary Outcome: Inner Macular Thickness (Inferior)
Description: Macular thickness was measured by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Week 12 (Day 85)
Population: Safety analysis set - Participants in the safety analysis set with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 24 | 28 | 31
micrometer | 503.06 (137.235) | 400.82 (53.180) | 390.48 (48.097)

7. Primary Outcome: Inner Macular Thickness (Temporal)
Description: Macular thickness was measured by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Week 12 (Day 85)
Population: Safety analysis set - Participants in the safety analysis set with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 24 | 28 | 31
micrometer | 505.27 (141.410) | 414.64 (67.032) | 404.93 (56.099)

8. Primary Outcome: Outer Macular Thickness (Inferior)
Description: Macular thickness was measured by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Week 12 (Day 85)
Population: Safety analysis set - Participants in the safety analysis set with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 23 | 28 | 31
micrometer | 388.66 (88.128) | 349.39 (44.538) | 342.88 (50.612)

9. Primary Outcome: Outer Macular Thickness (Temporal)
Description: Macular thickness was measured by spectral domain optical coherence tomography (SD-OCT).
Time Frame: Week 12 (Day 85)
Population: Safety analysis set - Participants in the safety analysis set with a valid measurement for the outcome measure.
Measure: Mean (Standard Deviation); unit: micrometer
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 23 | 28 | 31
micrometer | 404.60 (103.616) | 371.83 (70.124) | 352.24 (56.793)

10. Primary Outcome: Number of Participants Without Changes in Foveal Avascular Zone as Measured by Fluorescein Angiography (FA) in Study Eye
Description: Foveal avascular zone was assessed by fluorescein angiography (FA).
Time Frame: Days 29, 57, 85, End of Study (Up to Day 140)
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 21 | 25 | 30
Participants
  Day 29 - NO CHANGE: number analyzed (Participants) | 3 | 16 | 11
  Day 29 - NO CHANGE | 3 | 16 | 11
  Day 57 - NO CHANGE: number analyzed (Participants) | 3 | 16 | 7
  Day 57 - NO CHANGE | 3 | 16 | 7
  Day 85 - NO CHANGE: number analyzed (Participants) | 21 | 25 | 29
  Day 85 - NO CHANGE | 21 | 25 | 29
  End of Study (Up to Day 140) - NO CHANGE: number analyzed (Participants) | 17 | 23 | 30
  End of Study (Up to Day 140) - NO CHANGE | 17 | 22 | 30
  End of Study (Up to Day 140) - CANNOT GRADE: number analyzed (Participants) | 0 | 23 | 0
  End of Study (Up to Day 140) - CANNOT GRADE |  | 1 |

11. Primary Outcome: Mixed Model Repeated Measures Analysis of Ratio to Baseline in Central Subfield Retinal Thickness (CSFT) in the Study Eye
Description: Central subfield thickness was measured by spectral domain optical coherence tomography (SD-OCT). Central subfield retinal thickness was analyzed with a mixed model for repeated measures. The model included treatment, visit, and the treatment by visit interaction as independent variables. An unstructured residual covariance structure was used. Log-transformed baseline central subfield retinal thickness and treatment naïve and treatment experienced variable were used as covariates. Results were back-transformed to show results as a ratio to baseline.
Time Frame: Days 8, 15, 29, 43, 57, 85
Population: as for outcome 5
Measure: Geometric Mean (90% Confidence Interval); unit: ratio
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 25 | 28 | 32
ratio
  Day 8: number analyzed (Participants) | 6 | 16 | 10
  Day 8 | 0.99 [0.92 to 1.07] | 0.83 [0.78 to 0.88] | 0.83 [0.78 to 0.88]
  Day 15: number analyzed (Participants) | 6 | 16 | 10
  Day 15 | 0.97 [0.90 to 1.05] | 0.83 [0.78 to 0.88] | 0.80 [0.76 to 0.86]
  Day 29 | 1.00 [0.94 to 1.05] | 0.80 [0.76 to 0.85] | 0.82 [0.78 to 0.86]
  Day 43: number analyzed (Participants) | 5 | 16 | 8
  Day 43 | 1.04 [0.97 to 1.13] | 0.76 [0.71 to 0.81] | 0.79 [0.74 to 0.84]
  Day 57: number analyzed (Participants) | 24 | 27 | 30
  Day 57 | 0.95 [0.89 to 1.00] | 0.75 [0.70 to 0.80] | 0.80 [0.76 to 0.84]
  Day 85: number analyzed (Participants) | 23 | 27 | 31
  Day 85 | 0.97 [0.91 to 1.05] | 0.75 [0.70 to 0.80] | 0.78 [0.73 to 0.83]
Statistical Analysis 1: Comparison: LKA651 vs Lucentis; Day 8; Test type: Superiority; p = 0.998, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.20, 90% CI 2-sided [1.08 to 1.33] — Comparison of model-based mean estimates
Statistical Analysis 2: Comparison: LKA651 + Lucentis vs Lucentis; Day 8; Test type: Superiority; p = 0.527, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.00, 90% CI 2-sided [0.92 to 1.09] — Comparison of model-based mean estimates
Statistical Analysis 3: Comparison: LKA651 vs Lucentis; Day 15; Test type: Superiority; p = 0.999, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.21, 90% CI 2-sided [1.10 to 1.33] — Comparison of model-based mean estimates
Statistical Analysis 4: Comparison: LKA651 + Lucentis vs Lucentis; Day 15; Test type: Superiority; p = 0.716, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.03, 90% CI 2-sided [0.95 to 1.12] — Comparison of model-based mean estimates
Statistical Analysis 5: Comparison: LKA651 vs Lucentis; Day 29; Test type: Superiority; p = 1.000, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.21, 90% CI 2-sided [1.13 to 1.31] — Comparison of model-based mean estimates
Statistical Analysis 6: Comparison: LKA651 + Lucentis vs Lucentis; Day 29; Test type: Superiority; p = 0.281, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 0.98, 90% CI 2-sided [0.91 to 1.05] — Comparison of model-based mean estimates
Statistical Analysis 7: Comparison: LKA651 vs Lucentis; Day 43; Test type: Superiority; p = 1.000, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.32, 90% CI 2-sided [1.20 to 1.46] — Comparison of model-based mean estimates
Statistical Analysis 8: Comparison: LKA651 + Lucentis vs Lucentis; Day 43; Test type: Superiority; p = 0.200, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 0.96, 90% CI 2-sided [0.88 to 1.04] — Comparison of model-based mean estimates
Statistical Analysis 9: Comparison: LKA651 vs Lucentis; Day 57; Test type: Superiority; p = 1.000, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 1.18, 90% CI 2-sided [1.09 to 1.28] — Comparison of model-based mean estimates
Statistical Analysis 10: Comparison: LKA651 + Lucentis vs Lucentis; Day 57; Test type: Superiority; p = 0.083, Mixed model repeated measures analysis; Ratio (Test vs Reference) = 0.94, 90% CI 2-sided [0.87 to 1.01] — Comparison of model-based mean estimates
Statistical Analysis 11: Comparison: LKA651 vs Lucentis; Day 85; Test type: Superiority; p = 1.000, Mixed model repeated measures analysis; Ratio(Test vs Reference) = 1.26, 90% CI 2-sided [1.14 to 1.38] — Comparison of model-based mean estimates
Statistical Analysis 12: Comparison: LKA651 + Lucentis vs Lucentis; Day 85; Test type: Superiority; p = 0.254, Mixed model repeated measures analysis; Ratio(Test vs Reference) = 0.96, 90% CI 2-sided [0.88 to 1.06] — Comparison of model-based mean estimates

12. Secondary Outcome: Number of Participants Who Needed Retreatment With Anti-VEGF in Study Eye After Week 12
Time Frame: Week 12 (Day 85) up to Day 140
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 25 | 29 | 32
Participants | 16 | 16 | 21

13. Secondary Outcome: Time to Retreatment in Study Eye With Anti-VEGF After Week 12
Description: Time to retreatment with anti VEGF (as determined by the investigator) after Week 12 during the additional 12 week extension phase (that was up to 16 weeks after the last dose) was examined with a Kaplan Meier plot.
Time Frame: Week 12 (Day 85) up to Day 140
Population: as for outcome 5
Measure: Median (95% Confidence Interval); unit: Days after Day 85 (Week 12)
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 25 | 29 | 32
Days after Day 85 (Week 12) | 55.0 [17.0 to NA] — Not estimable due to insufficient number of participants with events. | 34.0 [12.0 to NA] — Not estimable due to insufficient number of participants with events. | 31.0 [9.0 to 109.0]

14. Secondary Outcome: Summary Statistics of Pharmacokinetics - Serum Concentrations of LKA651
Description: PK parameters were determined using non-compartmental methods using the most recent version of WinNonlin Phoenix (Version 8.2).
  Concentrations below the lower limit of quantification (LLOQ) were treated as 1/2 LLOQ in summary statistics.
Time Frame: Day 1 (0, 0.5 and 4 hrs post dose), Day 2, Day 8, Day 15, Day 29 (0, 0.5 and 4 hrs post dose), Day 43, Day 57 (0, 0.5 and 4 hrs post dose), Day 85
Population: Pharmacokinetic analysis set. Concentrations below the Lower Limit of Quantification (LLOQ) are reported as zero.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 23 | 28 | 0
ng/mL
  Day 1 - 0 hrs | 0.00 (0.00) | 0.00 (0.00) |
  Day 1 - 0.5 hrs post dose: number analyzed (Participants) | 1 | 8 | 0
  Day 1 - 0.5 hrs post dose | 0.00 | 0.00 (0.00) |
  Day 1 - 4 hrs post dose: number analyzed (Participants) | 6 | 15 | 0
  Day 1 - 4 hrs post dose | 114 (211) | 4.43 (17.1) |
  Day 2: number analyzed (Participants) | 6 | 15 | 0
  Day 2 | 36.3 (29.2) | 8.13 (21.6) |
  Day 8: number analyzed (Participants) | 6 | 15 | 0
  Day 8 | 16.2 (27.5) | 2.08 (8.06) |
  Day 15: number analyzed (Participants) | 5 | 15 | 0
  Day 15 | 7.24 (16.2) | 0.00 (0.00) |
  Day 29 - 0 hrs: number analyzed (Participants) | 22 | 24 | 0
  Day 29 - 0 hrs | 0.00 (0.00) | 0.00 (0.00) |
  Day 29 - 0.5 hrs post dose: number analyzed (Participants) | 1 | 6 | 0
  Day 29 - 0.5 hrs post dose | 0.00 | 0.00 (0.00) |
  Day 29 - 4 hrs post dose: number analyzed (Participants) | 0 | 6 | 0
  Day 29 - 4 hrs post dose |  | 7.60 (18.6) |
  Day 43: number analyzed (Participants) | 1 | 6 | 0
  Day 43 | 0.00 | 0.00 (0.00) |
  Day 57 - 0 hrs: number analyzed (Participants) | 21 | 23 | 0
  Day 57 - 0 hrs | 0.00 (0.00) | 0.00 (0.00) |
  Day 57 - 0.5 hrs post dos: number analyzed (Participants) | 1 | 6 | 0
  Day 57 - 0.5 hrs post dos | 0.00 | 0.00 (0.00) |
  Day 57 - 4 hrs post dose: number analyzed (Participants) | 0 | 6 | 0
  Day 57 - 4 hrs post dose |  | 0.00 (0.00) |
  Day 85: number analyzed (Participants) | 19 | 23 | 0
  Day 85 | 0.00 (0.00) | 0.00 (0.00) |

15. Secondary Outcome: Summary Statistics of Pharmacokinetics - AUC0-28d of LKA651 (Serum)
Description: Area under the curve over the dosing interval 0 to 28 days.
Time Frame: Day 1 - 4 hrs post dose, Day 2, Day 8, Day 15, Day 29 - 4 hrs post dose, Day 43, Day 57 - 4 hrs post dose, Day 85
Population: Pharmacokinetic analysis set. PK parameters could not be derived due to the limited number of LKA651 concentrations above the lower limit of quantification.
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 0 | 0 | 0

16. Secondary Outcome: Summary Statistics of Pharmacokinetics - Serum Concentrations of Lucentis
Time Frame: Day 1 - 4 hrs post dose, Day 2, Day 8, Day 15, Day 29 - 4 hrs post dose, Day 43, Day 57 - 4 hrs post dose, Day 85
Population: Pharmacokinetic analysis set. PK parameters could not be derived due to the limited number of Lucentis concentrations above the lower limit of quantification.
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 0 | 0 | 0

17. Secondary Outcome: Summary Statistics of Pharmacokinetics - AUC0-28d of Lucentis (Serum)
Description: Area under the curve over the dosing interval 0 to 28 days.
Time Frame: Day 1 - 4 hrs post dose, Day 2, Day 8, Day 15, Day 29 - 4 hrs post dose, Day 43, Day 57 - 4 hrs post dose, Day 85
Population: as for outcome 16
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 0 | 0 | 0

18. Post Hoc Outcome: All Collected Deaths
Description: On-treatment deaths are reported from first dose of study treatment until end of study treatment plus 12 weeks post treatment, up to a maximum timeframe of approximately 24 weeks (approximately 168 days).
  Post-treatment deaths are reported for the timeframe of greater than 30 days after last treatment, until study completion, up to approximately 168 days.
  All deaths refer to the sum of on-treatment and post-treatment deaths.
Time Frame: On-treatment - up to 12 weeks; Post-treatment - greater than 30 days after last treatment, until study completion, up to approximately 168 days
Population: Safety Set
Measure: Count of Participants; unit: Participants
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis
Number analyzed (Participants) | 28 | 30 | 33
Participants
  On-Treatment Deaths | 0 | 0 | 0
  Post-Treatment Deaths | 1 | 0 | 0
  All Deaths | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events are reported from first dose of study treatment until end of study treatment plus 12 weeks post treatment, up to a maximum timeframe of approximately 24 weeks (approximately 168 days).
Groups:
- Total: Total
Arm/Group | LKA651 | LKA651 + Lucentis | Lucentis | Total
All-Cause Mortality (participants affected / at risk) | 1/28 | 0/30 | 0/33 | 1/91
Serious Adverse Events (participants affected / at risk) | 3/28 | 4/30 | 1/33 | 8/91
Other Adverse Events (participants affected / at risk) | 20/28 | 16/30 | 19/33 | 55/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LKA651 (N=28) | LKA651 + Lucentis (N=30) | Lucentis (N=33) | Total (N=91)
Angina unstable (Cardiac disorders) | 0 | 1 | 0 | 1
Retinal detachment (Eye disorders) | 1 | 0 | 0 | 1
Cyclic vomiting syndrome (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Varices oesophageal (Gastrointestinal disorders) | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 1
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Bone cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | LKA651 (N=28) | LKA651 + Lucentis (N=30) | Lucentis (N=33) | Total (N=91)
Anaemia (Blood and lymphatic system disorders) | 1 | 2 | 1 | 4
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 1
Atrioventricular block first degree (Cardiac disorders) | 0 | 1 | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 0 | 1 | 1
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 1
Abnormal sensation in eye (Eye disorders) | 0 | 0 | 1 | 1
Anterior chamber flare (Eye disorders) | 0 | 1 | 0 | 1
Conjunctival haemorrhage (Eye disorders) | 1 | 5 | 2 | 8
Corneal erosion (Eye disorders) | 1 | 0 | 0 | 1
Cystoid macular oedema (Eye disorders) | 1 | 0 | 0 | 1
Dacryostenosis acquired (Eye disorders) | 1 | 0 | 0 | 1
Diabetic retinal oedema (Eye disorders) | 3 | 1 | 2 | 6
Diabetic retinopathy (Eye disorders) | 1 | 1 | 1 | 3
Dry eye (Eye disorders) | 0 | 1 | 1 | 2
Epiretinal membrane (Eye disorders) | 0 | 1 | 0 | 1
Eye pain (Eye disorders) | 1 | 0 | 0 | 1
Eyelids pruritus (Eye disorders) | 0 | 0 | 1 | 1
Lenticular opacities (Eye disorders) | 0 | 0 | 1 | 1
Macular oedema (Eye disorders) | 2 | 0 | 0 | 2
Ocular hypertension (Eye disorders) | 2 | 0 | 0 | 2
Punctate keratitis (Eye disorders) | 0 | 1 | 0 | 1
Retinal cyst (Eye disorders) | 1 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 1 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 1 | 0 | 0 | 1
Retinal oedema (Eye disorders) | 0 | 1 | 0 | 1
Visual acuity reduced (Eye disorders) | 3 | 0 | 0 | 3
Vitreoretinal traction syndrome (Eye disorders) | 0 | 0 | 1 | 1
Vitreous haemorrhage (Eye disorders) | 1 | 0 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hepatic steatosis (Hepatobiliary disorders) | 1 | 0 | 0 | 1
Hepatotoxicity (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Adenoviral conjunctivitis (Infections and infestations) | 0 | 1 | 1 | 2
COVID-19 (Infections and infestations) | 2 | 0 | 0 | 2
Conjunctivitis (Infections and infestations) | 1 | 0 | 0 | 1
Coronavirus infection (Infections and infestations) | 0 | 0 | 1 | 1
Herpes zoster (Infections and infestations) | 1 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 2
Sinusitis (Infections and infestations) | 0 | 2 | 0 | 2
Urinary tract infection (Infections and infestations) | 1 | 1 | 1 | 3
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
XIIth nerve injury (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 1
Blood cholesterol increased (Investigations) | 0 | 1 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 0 | 0 | 1
Blood creatinine increased (Investigations) | 2 | 0 | 0 | 2
Blood glucose increased (Investigations) | 1 | 1 | 0 | 2
Blood triglycerides increased (Investigations) | 1 | 0 | 1 | 2
Blood urea increased (Investigations) | 1 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 1 | 1
Glycosylated haemoglobin increased (Investigations) | 0 | 1 | 0 | 1
Intraocular pressure increased (Investigations) | 1 | 1 | 0 | 2
Lipase increased (Investigations) | 1 | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 1 | 0 | 1
Pancreatic enzymes increased (Investigations) | 1 | 0 | 0 | 1
Prostatic specific antigen increased (Investigations) | 0 | 1 | 0 | 1
SARS-CoV-2 test positive (Investigations) | 1 | 1 | 0 | 2
Urine ketone body present (Investigations) | 1 | 0 | 0 | 1
Urine leukocyte esterase positive (Investigations) | 1 | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Hypercholesterolaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 2 | 1 | 1 | 4
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperlipasaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 2 | 1 | 3
Vitamin B complex deficiency (Metabolism and nutrition disorders) | 0 | 1 | 0 | 1
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 2
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 1
Sjogren's syndrome (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 1 | 1
VIth nerve paralysis (Nervous system disorders) | 0 | 0 | 1 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 1 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0 | 1
Chronic kidney disease (Renal and urinary disorders) | 1 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0 | 1
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Essential hypertension (Vascular disorders) | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 3 | 1 | 3 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2022-07-06): https://cdn.clinicaltrials.gov/large-docs/90/NCT03927690/Prot_000.pdf
  • Statistical Analysis Plan (2022-08-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03927690/SAP_001.pdf